CLINICAL TRIAL: NCT01887015
Title: Early Nasal High Flow Oxygen Therapy for Prevention of Postoperative Hypoxemia After Abdominal Surgery: A Multicenter Randomized Controlled Trial
Brief Title: Optiflow® to Prevent Post-Extubation Hypoxemia afteR Abdominal Surgery (the OPERA Trial)
Acronym: OPERA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CHU-0157; 2013-A00030-45
Record Dates: First submitted 2013-06-24; First posted 2013-06-26 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Postoperative Hypoxemia
Keywords: Postoperative pulmonary complications; Oxygen therapy; Nasal high flow oxygen therapy; Nasal high flow cannula

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Standard oxygen therapy (Experimental): Our hypothesis is that, compared with standard oxygen therapy, early application of nasal high flow oxygen therapy can reduce the need for postoperative NPPV for postoperative hypoxemia (defined as PaO2/FiO2 ratio <300).
  Interventions: Device: Nasal high flow cannula (OptiflowTM, MR850 heated humidified, Fisher & Paykel Healthcare, Auckland, New Zealand)
- nasal high flow oxygen therapy (Other): Our hypothesis is that, compared with standard oxygen therapy, early application of nasal high flow oxygen therapy can reduce the need for postoperative NPPV for postoperative hypoxemia (defined as PaO2/FiO2 ratio <300).
  Interventions: Device: Nasal high flow cannula (OptiflowTM, MR850 heated humidified, Fisher & Paykel Healthcare, Auckland, New Zealand)

INTERVENTIONS:
Device: Nasal high flow cannula (OptiflowTM, MR850 heated humidified, Fisher & Paykel Healthcare, Auckland, New Zealand)
  Other Names: Nasal high flow oxygen therapy versus standard oxygen therapy

SUMMARY:
To evaluate whether early application of nasal high flow oxygen therapy after extubation can reduce the incidence of postoperative hypoxemia (defined as a PaO2/FiO2 ratio <300) after abdominal surgery in patients with intermediate to high risk of postoperative pulmonary complications.

DETAILED DESCRIPTION:
Postoperative hypoxemia complicates between 30 to 50% of patients after abdominal surgery. Loss of functioning alveolar units and development of atelectasis after abdominal surgery have been recognized as the underlying mechanisms responsible for postoperative hypoxemia. Supplemental Oxygen administration is therefore widely recommended after extubation in the postoperative period, especially in patients with high risk of postoperative respiratory complications. Although oxygen therapy is effective in preventing the vast majority of severe postoperative hypoxemia after extubation in surgical patients, respiratory failure may occur, thus requiring endotracheal intubation and mechanical ventilation or therapeutic use of non-invasive positive pressure ventilation (NPPV). In patients with postoperative hypoxemia (defined as patients with a PaO2/FiO2 ratio <300), application of NPPV was found to decrease the incidence of endotracheal intubation after abdominal surgery. Nevertheless, use of NPPV in the postoperative period is responsible for organizational constraints and increases healthcare utilization.

Nasal high flow cannula (NHFC) has been described as an attractive and well-tolerated method of non-invasive oxygen delivery. Previous studies have shown that NHFC generates a low level of positive airway pressure, increases end-expiratory lung volume and reduces airway resistance, thus contributing to a reduction in work of breathing. To date, however, no clinical trials have compared NHFC to standard oxygen therapy in the prevention of postoperative hypoxemia after abdominal surgery in patients with intermediate to high risk of postoperative pulmonary complications.

The primary objective of the study is to compare: 1- Standard oxygen therapy; 2- Nasal high flow oxygen therapy after extubation in patients with intermediate to high risk of postoperative pulmonary complications after abdominal surgery.

Our hypothesis is that, compared with standard oxygen therapy, early application of nasal high flow oxygen therapy can reduce the need for postoperative NPPV for postoperative hypoxemia (defined as PaO2/FiO2 ratio <300).

ELIGIBILITY:
Inclusion Criteria:

* Planned or unplanned surgical procedures
* Abdominal or abdominal and thoracic surgery
* Expected duration ≥2 hours
* ARISCAT score ≥26 points

Exclusion Criteria:

* Age <18 years
* Body mass index >35 kg/m2
* Sleep apnea syndrome
* Patient refusal
* Pregnancy and/or lactation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2013-06; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
percentage of patients who developed postoperative hypoxemia (defined as PaO2/FiO2 ratio <300) | 1 hour after tracheal extubation (day 1)

SECONDARY OUTCOMES:
Postoperative gas exchange (PaO2, PaCO2) | 1H after extubation and after surgery (at day 1)
Need for supplemental oxygen therapy beyond postoperative day 1 (defined as arterial oxygen saturation by pulse oximetry (SpO2) <93% in room air) | at day 1
Need for endotracheal intubation or non-invasive ventilation for postoperative acute respiratory failure (ARF) | within the first 7 days after surgery
  ARF (acute respiratory failure) is defined by one of the hypoxemic criteria (SpO2 <92% while breathing at least 10 L/min oxygen, PaO2 <60 mmHg on air or <80 mmHg while breathing any supplemental oxygen) and at least 1 of the following criteria: severe respiratory distress with dyspnea, accessory muscle recruitment and paradoxical abdominal or thoracic motion, respiratory rate >25 breaths/min, respiratory acidosis with pH <7.30 and PaCO2 > 50 mmHg.
Postoperative pulmonary complications (PPCs) | within the first 7 days after surgery
  PPCs(Postoperative pulmonary complications ) are scored using a grade scale ranging from 0 to 4, with grade 0 representing the absence of any complications and grade 1 through 4 representing successively the worse forms of complications.
Respiratory discomfort using a numerical rating scale (NRS) ranging from 0 (no discomfort) to 10 (maximum imaginable discomfort). | within the first 7 days after surgery
  Discomfort symptoms are assessed by evaluating dryness of the nose, mouth and throat.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel FUTIER, MD, Ph D, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Futier E, Paugam-Burtz C, Godet T, Khoy-Ear L, Rozencwajg S, Delay JM, Verzilli D, Dupuis J, Chanques G, Bazin JE, Constantin JM, Pereira B, Jaber S; OPERA study investigators. Effect of early postextubation high-flow nasal cannula vs conventional oxygen therapy on hypoxaemia in patients after major abdominal surgery: a French multicentre randomised controlled trial (OPERA). Intensive Care Med. 2016 Dec;42(12):1888-1898. doi: 10.1007/s00134-016-4594-y. Epub 2016 Oct 22. PMID 27771739
- [Derived] Futier E, Paugam-Burtz C, Constantin JM, Pereira B, Jaber S. The OPERA trial - comparison of early nasal high flow oxygen therapy with standard care for prevention of postoperative hypoxemia after abdominal surgery: study protocol for a multicenter randomized controlled trial. Trials. 2013 Oct 18;14:341. doi: 10.1186/1745-6215-14-341. PMID 24138710